CLINICAL TRIAL: NCT00850707
Title: Artero-venous Fistula, Prosthetic Polytetrafluoroethylene Grafts (AVG), Tunneled Cuffed Catheter (TCC): Impact of Vascular Access on HD Inflammation and Monocyte Activation
Brief Title: Vascular Access for Hemodialysis and Inflammation
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Prof.Sergio Stefoni, St.Orsola University Hospital
Other Study IDs: VASACC2009-02
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Vascular Access for Hemodialysis and Inflammation
Keywords: AVF; AVG; TCC; inflammation; monocite senescence
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: 220 hemodialysis patients with Arterovenous fistula (AVF group)
- 2: 58 hemodialysis patients with Arterovenous graft (AVG group)
- 3: 180 hemodialysis patients with Tunneled cuffed catheters (TCC group)
- 4: 60 healthy subjects as controls

SUMMARY:
The aim of the present study was to investigate patients free of active infection and/or thrombosis to assess if the type of vascular access (AVF, AVG, TCC), could influence:

1. the levels of serological markers of inflammation (CRP, IL-6, TNF-a);
2. the degree of expression on monocyte surface of inflammation and immune response modulating molecules: CD14, CD32 and CD44.
3. the amount of monocytic cells expressing a senescent phenotype (CD14 and CD32).

DETAILED DESCRIPTION:
Patients with AVF assumed ticlopidine 250 mg/die, patients with TCC and AVG assumed warfarin to maintain target INR between 1.8 and 2.5.

Six wash out consecutive sessions were carried out before starting the study with Fresenius FX8 Helyxone® , for patients who underwent HD, or with FX 80 Helyxone®, for patients who underwent hemodiafiltration (HDF). After the wash out period, fresh whole blood and serum samples were drawn on starting dialysis, during the midweek HD session for 4 consecutive weeks. For each patient the mean value of the 4 blood samples was considered. All patients continued HD or HDF with FX8 or FX 80 Helyxone® during the whole study period.In order to estimate the normal ranges of the parameters that we evaluated, 60 anonymous healthy volunteers were also submitted to the same assays.

ELIGIBILITY:
Inclusion Criteria:

* All the patients recruited for the study were infection and thrombosis free from almost 6 months.
* No patients included had autoimmune disease, hepatic failure, diabetes or malignancy.
* Patients were not administered ACE inhibitors, angiotensin receptor antagonists, antiinflammatory or immunosuppressive drugs.
* All the patients had residual GFR < 5 ml/min.
* The vascular access considered were placed from at least 6 months.

Exclusion Criteria:

* Patients with recirculating vascular access > 10% were excluded from the study.
* Patients with acute cardiovascular accident in the last 15 days before starting the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The three groups of patients were homogeneous for: a) demographic characteristics; b) dialysis adequacy; c) vascular access blood flow; d) white cell count.
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2000-01; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
serological markers of inflammation (CRP, IL-6, TNF-a) | 6 weeks
monocyte surface of inflammation and immune response modulating molecules: CD14, CD32 and CD44. | 6 weeks
monocytic cells expressing a senescent phenotype (CD14 and CD32). | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Dialysis Transplantation Unit St.Orsola University Hospital, Bologna, Italy

REFERENCES:
- [Background] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Background] Weiss MF, Scivittaro V, Anderson JM. Oxidative stress and increased expression of growth factors in lesions of failed hemodialysis access. Am J Kidney Dis. 2001 May;37(5):970-80. doi: 10.1016/s0272-6386(05)80013-7. PMID 11325679
- [Background] Nilsson B, Ekdahl KN, Mollnes TE, Lambris JD. The role of complement in biomaterial-induced inflammation. Mol Immunol. 2007 Jan;44(1-3):82-94. doi: 10.1016/j.molimm.2006.06.020. Epub 2006 Aug 14. PMID 16905192
- [Background] Bologa RM, Levine DM, Parker TS, Cheigh JS, Serur D, Stenzel KH, Rubin AL. Interleukin-6 predicts hypoalbuminemia, hypocholesterolemia, and mortality in hemodialysis patients. Am J Kidney Dis. 1998 Jul;32(1):107-14. doi: 10.1053/ajkd.1998.v32.pm9669431.
- [Background] Zimmermann J, Herrlinger S, Pruy A, Metzger T, Wanner C. Inflammation enhances cardiovascular risk and mortality in hemodialysis patients. Kidney Int. 1999 Feb;55(2):648-58. doi: 10.1046/j.1523-1755.1999.00273.x. PMID 9987089
- [Background] Yeun JY, Levine RA, Mantadilok V, Kaysen GA. C-Reactive protein predicts all-cause and cardiovascular mortality in hemodialysis patients. Am J Kidney Dis. 2000 Mar;35(3):469-76. doi: 10.1016/s0272-6386(00)70200-9. PMID 10692273
- [Background] Ramirez R, Carracedo J, Soriano S, Jimenez R, Martin-Malo A, Rodriguez M, Blasco M, Aljama P. Stress-induced premature senescence in mononuclear cells from patients on long-term hemodialysis. Am J Kidney Dis. 2005 Feb;45(2):353-9. doi: 10.1053/j.ajkd.2004.10.022. PMID 15685514
- [Background] Carracedo J, Ramirez R, Madueno JA, Soriano S, Rodriguez-Benot A, Rodriguez M, Martin-Malo A, Aljama P. Cell apoptosis and hemodialysis-induced inflammation. Kidney Int Suppl. 2002 May;(80):89-93. doi: 10.1046/j.1523-1755.61.s80.17.x. PMID 11982820
- [Background] Kielian TL, Blecha F. CD14 and other recognition molecules for lipopolysaccharide: a review. Immunopharmacology. 1995 Apr;29(3):187-205. doi: 10.1016/0162-3109(95)00003-c. PMID 7542643
- [Background] Patino R, Ibarra J, Rodriguez A, Yague MR, Pintor E, Fernandez-Cruz A, Figueredo A. Circulating monocytes in patients with diabetes mellitus, arterial disease, and increased CD14 expression. Am J Cardiol. 2000 Jun 1;85(11):1288-91. doi: 10.1016/s0002-9149(00)00757-8. PMID 10831941
- [Background] Ramirez R, Carracedo J, Berdud I, Carretero D, Merino A, Rodriguez M, Tetta C, Martin-Malo A, Aljama P. Microinflammation in hemodialysis is related to a preactivated subset of monocytes. Hemodial Int. 2006 Jan;10 Suppl 1:S24-7. doi: 10.1111/j.1542-4758.2006.01186.x. PMID 16441864
- [Background] Tacke F, Randolph GJ. Migratory fate and differentiation of blood monocyte subsets. Immunobiology. 2006;211(6-8):609-18. doi: 10.1016/j.imbio.2006.05.025. Epub 2006 Jul 10. PMID 16920499
- [Background] Pure E, Cuff CA. A crucial role for CD44 in inflammation. Trends Mol Med. 2001 May;7(5):213-21. doi: 10.1016/s1471-4914(01)01963-3. PMID 11325633
- [Background] Gee K, Lim W, Ma W, Nandan D, Diaz-Mitoma F, Kozlowski M, Kumar A. Differential regulation of CD44 expression by lipopolysaccharide (LPS) and TNF-alpha in human monocytic cells: distinct involvement of c-Jun N-terminal kinase in LPS-induced CD44 expression. J Immunol. 2002 Nov 15;169(10):5660-72. doi: 10.4049/jimmunol.169.10.5660. PMID 12421945
- [Background] Movilli E, Brunori G, Camerini C, Vizzardi V, Gaggia P, Cassamali S, Scolari F, Parrinello G, Cancarini GC. The kind of vascular access influences the baseline inflammatory status and epoetin response in chronic hemodialysis patients. Blood Purif. 2006;24(4):387-93. doi: 10.1159/000093681. Epub 2006 Jun 1. PMID 16755161
- [Background] Chang CJ, Ko YS, Ko PJ, Hsu LA, Chen CF, Yang CW, Hsu TS, Pang JH. Thrombosed arteriovenous fistula for hemodialysis access is characterized by a marked inflammatory activity. Kidney Int. 2005 Sep;68(3):1312-9. doi: 10.1111/j.1523-1755.2005.00529.x. PMID 16105066
- [Background] Raad I, Costerton W, Sabharwal U, Sacilowski M, Anaissie E, Bodey GP. Ultrastructural analysis of indwelling vascular catheters: a quantitative relationship between luminal colonization and duration of placement. J Infect Dis. 1993 Aug;168(2):400-7. doi: 10.1093/infdis/168.2.400. PMID 8335977
- [Background] Beathard GA, Urbanes A. Infection associated with tunneled hemodialysis catheters. Semin Dial. 2008 Nov-Dec;21(6):528-38. doi: 10.1111/j.1525-139X.2008.00497.x. Epub 2008 Sep 24. PMID 19000122
- [Background] Kaysen GA. The microinflammatory state in uremia: causes and potential consequences. J Am Soc Nephrol. 2001 Jul;12(7):1549-1557. doi: 10.1681/ASN.V1271549. PMID 11423586
- [Background] Ayus JC, Sheikh-Hamad D. Silent infection in clotted hemodialysis access grafts. J Am Soc Nephrol. 1998 Jul;9(7):1314-7. doi: 10.1681/ASN.V971314. PMID 9644644
- [Background] Roy-Chaudhury P, Kelly BS, Miller MA, Reaves A, Armstrong J, Nanayakkara N, Heffelfinger SC. Venous neointimal hyperplasia in polytetrafluoroethylene dialysis grafts. Kidney Int. 2001 Jun;59(6):2325-34. doi: 10.1046/j.1523-1755.2001.00750.x. PMID 11380837
- [Background] Oliver MJ, Mendelssohn DC, Quinn RR, Richardson EP, Rajan DK, Pugash RA, Hiller JA, Kiss AJ, Lok CE. Catheter patency and function after catheter sheath disruption: a pilot study. Clin J Am Soc Nephrol. 2007 Nov;2(6):1201-6. doi: 10.2215/CJN.01910507. Epub 2007 Oct 17. PMID 17942775
- [Background] Daneshian M, Wendel A, Hartung T, von Aulock S. High sensitivity pyrogen testing in water and dialysis solutions. J Immunol Methods. 2008 Jul 20;336(1):64-70. doi: 10.1016/j.jim.2008.03.013. Epub 2008 Apr 24. PMID 18474369